CLINICAL TRIAL: NCT06532747
Title: Redefining BMI: The Body, Mind, and Inflammation Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HM20028726
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Adiposity
Keywords: BMI; Emerging Adult (EA) Women; Lifestyle Intervention; Biomarker Inflammation Improvement
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This is a 2-arm, parallel randomized controlled pilot trial designed to test the preliminary efficacy of a novel integrated lifestyle intervention for emerging adult (EA) women, compared to a developmentally adapted behavioral weight loss arm.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Lifestyle Intervention (ILI) (Experimental): ILI participants will receive training in empirically supported strategies to improve psychological function (e.g., restructuring negative thoughts, distress tolerance), with a focus on changing discrete behaviors linked to inflammation (e.g., sleep, processed foods, physical activity), all intertwined with BWL content adapted to meet the needs of EAs.
  All participants will receive digital tools to facilitate self-monitoring-the initial 4-month program will consist of group sessions via Zoom (8 weekly, 4 bi-weekly) with weekly tailored e-coaching, followed by monthly boosters through 12 months.
  Interventions: Behavioral: Integrated Lifestyle Intervention (ILI)
- Behavioral Weight Loss (BWL) (Experimental): All participants will receive digital tools to facilitate self-monitoring-the initial 4-month program will consist of group sessions via Zoom (8 weekly, 4 bi-weekly) with weekly tailored e-coaching, followed by monthly boosters through 12 months.
  Interventions: Behavioral: Integrated Lifestyle Intervention (ILI); Behavioral: Monitoring with digital tools

INTERVENTIONS:
Behavioral: Integrated Lifestyle Intervention (ILI) — ILI participants will receive training in empirically supported strategies to improve psychological function (e.g., restructuring negative thoughts, distress tolerance), with a focus on changing discrete behaviors linked to inflammation (e.g., sleep, processed foods, physical activity), all intertwined with BWL content adapted to meet the needs of EAs.
Behavioral: Monitoring with digital tools — All participants will receive digital tools to facilitate self-monitoring-the initial 4-month program will consist of group sessions via Zoom (8 weekly, 4 bi-weekly) with weekly tailored e-coaching, followed by monthly boosters through 12 months.
  Arms: Behavioral Weight Loss (BWL)

SUMMARY:
Emerging adulthood (18-25 years of age) is a critical developmental window to promote weight management and cardiometabolic health, particularly for emerging adult women. The primary purpose of this study is to test the preliminary efficacy of the intensive lifestyle intervention for EA women in reducing adiposity, as well as improving biomarkers of inflammation and metabolic risk over 12 months compared with a traditional behavioral weight loss intervention. This treatment program will be tested in emerging adult (EA) women ages 18-25 years old with a BMI of 25-50 kg/m^2.

DETAILED DESCRIPTION:
This is a 2-arm, parallel randomized controlled pilot trial designed to test the preliminary efficacy of a novel integrated lifestyle intervention for emerging adult (EA) women, compared to a developmentally adapted behavioral weight loss arm. Thirty-two participants (female, 18-25 years, BMI 25-50 kg/m^2) will be randomized to 1 of 2 arms: 1) Integrated Lifestyle Intervention (ILI); or 2) Behavioral Weight Loss (BWL). The primary goals are to test the preliminary efficacy of ILI to reduce adiposity over 12 months compared to BWL, and to test the preliminary efficacy of ILI to improve biomarkers of inflammation and cardiometabolic risk over 12 months compared with BWL. Assessments of adiposity, inflammatory cytokines, cardiovascular disease (CVD) risk factors, and behavioral and psychological treatment targets will occur at 0, 4, 8 and 12 months. In addition, putative psychological mechanisms of action will be explored to inform a future trial.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-25 years
* Body mass index (BMI) 25-50 kg/m^2
* Female

Exclusion Criteria:

* Currently pregnant or lactating
* Current involvement in a weight loss program or current use of weight loss medication
* Lost >5% of their body weight in the previous 3 months
* Uncontrolled medical conditions that may pose a safety issue given the recommendations for the diet and unsupervised physical activity
* Diagnosis of type 2 diabetes and/or impaired fasting blood glucose
* Diagnosis of type 1 diabetes
* Rheumatologic and gastrointestinal conditions associated with severe systemic inflammation
* Medical conditions resulting in known perturbations in the hypothalamic-pituitary-adrenal axis
* Report of a heart condition, chest pain during periods of activity or rest, or loss of consciousness
* Current or recent (during the past 3 months) use of medications that may impact weight or metabolic function
* Current or recent (during the past 3 months) use of anti-inflammatory medications
* Report of diagnosis or history of Anorexia Nervosa or Bulimia Nervosa, or any compensatory behaviors within the previous 3 months
* Hospitalization for depression or other psychiatric disorder within the past 12 months
* Uncontrolled bipolar disorder or psychotic disorder
* Current suicidal intent
* Planning to move from the area within the study period
* Unwilling to be randomized to either study condition
* Unable to read and speak English

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2027-03-03 (Estimated); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
To test the preliminary efficacy of the intensive lifestyle intervention for EA women in reducing adiposity over 12 months compared with BWL | Change in weight at 4, 8, and 12-months
  Change in adiposity (weight) between the two treatment arms across 12-months
To test the preliminary efficacy of the intensive lifestyle intervention for EA women in reducing waist circumference over 12 months compared with BWL | Change in waist circumference at 4, 8, and 12-months.
  Change in adiposity (waist circumference) between the two treatment arms across 12-months
To test the preliminary efficacy of the intensive lifestyle intervention for EA women in reducing % body fat over 12 months compared with BWL | Change in % body fat at 4, 8, and 12-months.
  Change in adiposity (% body fat) between the two treatment arms across 12-months

SECONDARY OUTCOMES:
To test the preliminary efficacy of ILI to improve biomarkers of inflammation and cardiometabolic risk over 12 months compared with BWL examining Change in serum IL-1β and IL-6 at 4, 8, and 12-months. | 4, 8, and 12-months
  Change in serum IL-1β and IL-6. Bursts of IL-1β can indicate acute inflammation, myocardial infarction, or stroke. IL-1β can also trigger the expression of IL-6 in various cell types. Elevated IL-6 levels can indicate an inflammatory condition, such as rheumatoid arthritis, lupus, or other autoimmune disorders. IL-6 levels can also correlate with disease activity.
To test the preliminary efficacy of ILI to improve biomarkers of inflammation and cardiometabolic risk over 12 months compared with BWL examining Change in serum TNF-α at 4, 8, and 12-months. | 4, 8, and 12-months
  Change in serum TNF-α. A systematic review and meta-analysis found that patients with T1DM had significantly higher serum TNF-α levels than controls. TNF-α levels were also correlated with age, disease duration, and ethnicity.
To test the preliminary efficacy of ILI to improve biomarkers of inflammation and cardiometabolic risk over 12 months compared with BWL examining Change in CRP at 4, 8, and 12-months. | 4, 8, and 12-months
  Change in CRP. Factors that can cause CRP levels to be slightly higher than normal include obesity, lack of exercise, cigarette smoking, diabetes, cancer, heart attack, inflammatory bowel disease (IBD), rheumatoid arthritis, lupus, and related diseases, and rheumatic fever.
To test the preliminary efficacy of ILI to improve biomarkers of inflammation and cardiometabolic risk over 12 months compared with BWL examining Change in free cortisol at 4, 8, and 12-months. | 4, 8, and 12-months
  Change in free cortisol, The normal range for adults is 3.5-45 micrograms per 24 hours, but this can vary by age. Factors that can affect free cortisol levels include: Stress, Alcoholism, Depression.
To test the preliminary efficacy of ILI to improve biomarkers of inflammation and cardiometabolic risk over 12 months compared with BWL examining Change in HOMA-IR at 4, 8, and 12-months | 4, 8, and 12-months
  Change in HOMA-IR, HOMA-IR measures the insulin level needed in the blood to maintain normal sugar levels. This test helps diagnose insulin resistance, the early stage of type 2 diabetes, a condition that increases the risks of several chronic health conditions.
Change in cholesterol level at 4, 8, and 12-months. | 4, 8, and 12-months
  Change in lipids, Lipid disorders can lead to serious health problems, such as heart disease and stroke, because they prevent the body from properly metabolizing fats. High levels of certain lipids, especially cholesterol, can also lead to long-term problems like atherosclerosis.
To test the preliminary efficacy of ILI to improve biomarkers of inflammation and cardiometabolic risk over 12 months compared with BWL examining Change in ALT/AST at 4, 8, and 12-months. | 4, 8, and 12-months
  Change in ALT/AST (Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)) There are many causes of mildly elevated ALT and AST levels. The most common causes are nonalcoholic fatty liver disease (NAFLD) and alcoholic liver disease. In NAFLD, the liver has more fatty tissue in it than normal.
To test the preliminary efficacy of ILI to improve biomarkers of inflammation and cardiometabolic risk over 12 months compared with BWL examining Change in systolic and diastolic blood pressure at 4, 8, and 12-months. | 4, 8, and 12-months
  Change in systolic and diastolic blood pressure. Your systolic and diastolic pressures change depending on your activity level, stress, fluid intake, and other factors. It's important to limit how these other factors might change your pressure when you're taking a blood pressure reading.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica LaRose, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth Universtity, Richmond, Virginia, United States